CLINICAL TRIAL: NCT05644704
Title: SportSense 6D Fusion - Application of Multi-sensor Fusion Environment in Movement, Training and Injury Prevention in Bat and Arm Swing Sports-Intelligent Sports Injury Prevention and Training System
Brief Title: Intelligent Sports Injury Prevention and Training System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202210101RIND
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Sport Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baseball pitcher training (Experimental)
  Interventions: Other: Lower extremity and core muscle training

INTERVENTIONS:
Other: Lower extremity and core muscle training — Lower extremity training: single leg balance training Core muscle training: pelvic control training

SUMMARY:
Sports injuries are a very important issue for baseball players. Previous studies have found that the incidence of sports injuries faced by baseball players is continuously increasing. Sports injury rates in professional baseball, high school baseball, and college baseball players were as high as 3.6, 4.6, and 5.8 per 1,000 players, respectively. The main cause of many pitching injuries is attributed to a large number of repetitive pitches. To avoid sports injuries, it is necessary to know how to assess the risk of injury caused by repetitive pitching. Throwing is a fairly complex action that requires the coordination of the entire body. It is critical to investigate the biomechanical changes of players in order to effectively analyze such complex movements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy baseball pitchers
* Age between 18~55 years old

Exclusion Criteria:

* Surgery history in pitching arm
* Musculoskeletal disease
* Neuromuscular disease

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-12 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Countermovement jump (CMJ) | 6 weeks
  Test CMJ before and after training

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang SM, Chen SH, Chen HY, Huang JH, Wu YR, Hsu WL. Pelvic Control and Pelvic-Trunk Coordination as Key Determinants of Pitching Velocity in Baseball Pitchers. Orthop J Sports Med. 2025 Jul 24;13(7):23259671251350302. doi: 10.1177/23259671251350302. eCollection 2025 Jul. PMID 40727237